CLINICAL TRIAL: NCT06325228
Title: Incidence and Relationshipis of Musculoskeletal Injuries, Sports Performance, Sports Specialization, and Quality of Life in Young Athletes. Project: "Science of Healthy Sport"
Brief Title: Musculoskeletal Injuries, Sports Performance, Sports Specialization, and Quality of Life in Young Athletes
Status: Completed | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Collaborators: Ministry of Science and Higher Education, Poland (Other Government)
Responsible Party: Principal Investigator, Bartosz Wilczyński, Principal Investigator, Medical University of Gdansk
Other Study IDs: NKBBN/241/2023; SONP/SP/549693/2022 (Other Grant/Funding Number: Minister of Education and Science)
Record Dates: First submitted 2024-03-10; First posted 2024-03-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Sport Injury; Healthy; Injury;Sports; Quality of Life
Keywords: Sports specialization; Young Athletes; Injury prevention; Sports performance
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young Athletes: 300 young athletes (boys and girls, 9 - 16 years-old) from clubs, teams, associations, sports classes of various disciplines in the Pomeranian Voivodeship

SUMMARY:
The primary aim of this observational cohort study is to assess sports specialization, sports performance, history of injuries (prevalence, types, areas, duration) and quality of life in young healthy athletes aged 8-16 from Poland. Athlete profiles will be created based on the variables (explained in detailed description) examined. Furthermore, the investigators will perform one-year injury follow-up.

The main questions it aims to answer are:

* Do athletes with a specific profile (lower values in athletic performance tests, low values in quality of life) evaluated at one time point, suffer injury in the future in annual observation?
* Do athletes with high sports specialization will sustain injury in one-year follow-up?
* Does sports specialization have a relationship with sports performance tests, and quality of life?
* Does sport specialisation, training volume, geographical factor relate to injury history?
* Does sports specialisation, injury history differ between sports (individual and team sports)?
* Does value of the specific muscle (lower limb) isometric strength will be associated with the dynamic balance scores in young healthy athletes?

DETAILED DESCRIPTION:
Recruited young healthy athletes (8-16 years-old) from sports schools, clubs, teams will invited to study. There will be performed assessment, which included:

* participant characteristics (age, biological age, gender, height, weight, body mass index, sports experience, training workload, sports specialization, history of injuries)
* sports performance (value of dynamic balance, isometric strength of lower limbs, functional movement patterns)
* quality of life and health assessment (EQ-5D-Y)
* geographical factor (Rural, Urban)
* Sports (Individual, Team)
* History of Injuries (Localization, Type)

One-year after meetings, there will be send questionaire and phone-call to participants and their coaches/parents in order to obtain information about injuries (location, type, time-loss, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Healthy (without injury, pain, or symptoms)
* Participation in sports activities (minimum 6 months)
* Age of 8 to 16 years-old
* Agreement to participation from parent/guardian

Exclusion Criteria:

* pain or other symptoms related during study
* lower extremity or trunk surgery in the last 6 months
* lack of medical approval for participation in sports games

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Young healthy athletes (8-16 years-old) from sports schools, clubs, teams from the territory of the Pomeranian voivodeship, Poland.
Sampling Method: Non-Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with sports injury after one-year follow-up | One year after the date of examination
  Dichotomous assessment (0 = no injury, 1 = injury) based on a telephone interview with the parent/guardian/coach. Conditions to meet: 12 months after the date of examination, and continuity of participation in sports to the date of injury
Type, location, duration, and return to sports in participants with injury at one-year follow up | One year after the date of examination
  Assessment based on a telephone interview with the parent/guardian/coach.
  Questions about:
  * exact type of injury (acute or chronic, contact or non-contact)
  * location of injury (anatomic site, e.g. knee)
  * duration of injury (time-loss, in days)
  * return to sports (Does the participant return to sport, yes or no)

SECONDARY OUTCOMES:
Sports Specialization | through study completion, an average of 1 year
  Sports specialization defined as "intensive year-round training in a single sport at the exclusion of other sports". Where a highly specialized athlete may be able to (1) choose a main sport, (2) participate for greater than 8 months per year in 1 main sport, and (3) quit all other sports to focus on 1 sport.
History of sports-related injuries | through study completion, an average of 1 year
  Questionaire - Question about sports-related injuries within sports career (sports participating in trainings and competitions) which included:
  * - exact type of injury (acute or chronic, contact or non-contact)
  * location of injury (anatomic site, e.g. knee)
  * duration of injury (time-loss, in days)
  Answers will be performed from young athlete and coach. If there will be occasion, answers will be matched with answers from parents/guardians.
Health-related quality of life: EQ-5D-Y | through study completion, an average of 1 year
  Patient Reported Outcome instruments" EQ-5D-Y - EuroQol Research Foundation - Certified Translation: Polish for Poland. The EQ-5D is a widely used standardized generic measure of HRQOL. A valid and accurate translation of the corresponding original document. A child-friendly version of the EQ-5D (0-100 points, where "0" means the worse quality of life, and "100" means perfect). (EQ-5D is the name of the instrument and is not an acronym.)
Y-Balance Test - dynamic balance test | through study completion, an average of 1 year
  Dynamic Balance of the lower extremities (record as reach distance in centimeters "cm" and normalized reach distance in percentages "%")
Functional Movement Screen (FMS) | through study completion, an average of 1 year
  The Functional Movement Screen (FMS) is a screening tool used to identify limitations or asymmetries in movement patterns. FMS consists of 7 movement tasks (deep squat, lunges, hurdle steps, a push-up, straight-leg raises, shoulder mobility, and rotary stability). Each task will be visually assessed by an experienced physiotherapist and marked on a 4-point scale (0-3, worst-best). The total maximum score that can be obtained is 21 points.
Hand-Held Dynamometer (HHD) measurement - Isometric Strength of the lower extremities muscle | through study completion, an average of 1 year
  Hand-Held Dynamometer (HHD) measurement (Laffayette, USA). Isometric Strength (peak force, average force (kilograms), of the lower extremities muscle (gluteus medium, quadriceps, hamstring, triceps surae.

OTHER OUTCOMES:
Sport workload (hours per trainings or competition) | through study completion, an average of 1 year
  Sports and training volume (hours per trainings or competition, weekly)
Peak Height Velocity | through study completion, an average of 1 year
  Peak Height Velocity (PHV) calculated using the 'maturity offset' value (report as "PHV years") - Mirwald formula
Sports discipline and position | through study completion, an average of 1 year
  Sport discipline (e.g. soccer) and Sports position (e.g. on the soccer field: defender)
Participants characteristics - Body Mass Index | through study completion, an average of 1 year
  weight and height will be combined to report BMI in kg/m^2
Sports experience | through study completion, an average of 1 year
  Sports experience (years, months)

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz Wilczyński, phD, Principal Investigator — Department of Immunobiology and Environment Microbiology, Medical University of Gdańsk
Locations (1):
- Department of Immunobiology and Environment Microbiology, Medical University of Gdańsk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
  The data that will be collected include data sets, i.e., personal survey questionnaires, measurement scales, functional and anthropometric assessment measurements, described in the description section of the scientific activity.
  Part of the data will be published in the public repository of the Polish Medical Research Platform and the Zenodo repository. Part of the data will be published in scientific journals, which may also require publication of raw data. Data will be made available at the latest at the time of publication.
  Data are available indefinitely at Polish Medical Research Platform and the Zenodo repository.
Supporting Information: Study Protocol, CSR
Time Frame: Immediately following publication. No end date
Access Criteria: Anyone who wishes to access the data

REFERENCES:
- [Background] Wilczynski B, Radziminski L, Sobierajska-Rek A, de Tillier K, Bracha J, Zorena K. Biological Maturation Predicts Dynamic Balance and Lower Limb Power in Young Football Players. Biology (Basel). 2022 Aug 3;11(8):1167. doi: 10.3390/biology11081167. PMID 36009793
- [Background] Wilczynski B, Radziminski L, Sobierajska-Rek A, Zorena K. Association between Selected Screening Tests and Knee Alignment in Single-Leg Tasks among Young Football Players. Int J Environ Res Public Health. 2022 May 31;19(11):6719. doi: 10.3390/ijerph19116719. PMID 35682301
- [Background] Bruzda R, Wilczynski B, Zorena K. Knee function and quality of life in adolescent soccer players with Osgood Shlatter disease history: a preliminary study. Sci Rep. 2023 Nov 6;13(1):19200. doi: 10.1038/s41598-023-46537-7. PMID 37932373
- [Background] Wilczynski B, Hinca J, Slezak D, Zorena K. The Relationship between Dynamic Balance and Jumping Tests among Adolescent Amateur Rugby Players. A Preliminary Study. Int J Environ Res Public Health. 2021 Jan 4;18(1):312. doi: 10.3390/ijerph18010312. PMID 33406658
- [Derived] Wilczynski B, Buler J, Buler RL, Grochowski ML, Puchalski B, Zorena K. Strength and balance asymmetries in children and adolescents: comparison between single- and multi-sport participants. BMC Sports Sci Med Rehabil. 2025 Nov 27;17(1):358. doi: 10.1186/s13102-025-01420-y. PMID 41310813

DOCUMENTS (1):
  • Informed Consent Form (2023-01-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT06325228/ICF_000.pdf